CLINICAL TRIAL: NCT03480425
Title: Force of Endotracheal Tube Extubation; Esophagus vs. Trachea; an Exploratory Crossover Clinical Trial
Brief Title: Force of Endotracheal Tube Extubation; Esophagus vs. Trachea
Acronym: TETT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analysis of first 10 participants showed the technique was not efficacious
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, Professor Emeritus, University of Saskatchewan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Bio# 17-273
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Esophageal then tracheal intubated patient (Experimental): Esophagus is intentionally intubated with a cuffed endotracheal tube, the cuff inflated to >30cm water pressure, a force transducer attached, and force of extubation recorded. Then Trachea is intentionally intubated the cuff inflated to >30cm water pressure, and force of extubation recorded.
  Interventions: Diagnostic Test: Measuring extubation force

INTERVENTIONS:
Diagnostic Test: Measuring extubation force — Intubation of the esophagus of anesthetized participants who are having planned endotracheal intubate for surgery; inflation of the cuff; attachment of a force transducer to the tube connector; and gently tugging the tube out of the mouth. Then intubating the esophagus and repeating the tugging procedure. Meanwhile, the force of resistance to tugging is measured with a force transducer.

SUMMARY:
A study of a new approach to determining if, following endotracheal intubation, the endotracheal tube (ETT) is in the trachea or the esophagus. The test for correct placement consists of inflating the cuff to a pressure of 50 (to be determined by the study) and tugging the ETT gently up and out of the mouth. The investigators hypothesize that if it is in the esophagus, it will slide easily all the way out; if in the trachea, the cuff will be impeded by catching on the lower surface of the cricoid ring, and that this will require a greater force to extubate with cuff inflated than that required for the esophagus.

DETAILED DESCRIPTION:
Correct endotracheal tube (ETT) placement is important. Ideal ETT position is achieved when the distal tip is in mid-trachea with the head in neutral alignment. Unrecognized tube misplacement is an uncommon but significant cause of hypoxemia and death during general anesthesia and emergency intubation of critically ill patients. It is commoner in out-of-hospital intubations, where it is reported to occur in 1 to 15% of cases, often with disastrous results. 1, 2 Three types of malpositioning can occur: one outside the trachea (esophageal), and two within the trachea: too shallow (hypopharyngeal), or too deep (endobronchial). Esophageal intubation results in rapid hypoxemia, hypercarbia, and inflation of the stomach as the patient receives no ventilation at all. 3 Too-shallow placement of the ETT can result in inadvertent extubation, especially with manipulation of head and neck. 4 Endobronchial intubation occurs when the ETT is advanced into a mainstem bronchus, which results in hypoxia and the potential for barotrauma in the hyperventilated lung. 5, 6 Confirmation of correct ETT depth is currently performed by several methods. In the operating room, simple measurement of the length of the tube at the corner of the mouth is rapid but not reliable. One study improved on this by using additional anatomical landmarks to determine ETT tube length as measured at the mouth.7 It enabled a reduction in the incidence of too-deep placement of the ETT from 58.8% to 24%.

Cuff ballottement at the level of the suprasternal notch is a technique that has been studied with cuffed tubes in adults. Ballottement as described in these papers involves moving the fingers in a direction normal to the long axis of the ETT in order to alternately compress and release the finger pressure on the cuff, while feeling and watching the corresponding movement of the pilot balloon. Ease of palpation of ballottement was inconsistent, and in one study 15 of 82 patients had ETT tips <2.5 cm above the carina. 8-10 Studies to date of ballottement do not comment on its ability to prevent esophageal intubation. Ultrasound guided intubation has been shown to provide correct placement, but requires training and machine availability. 11-14 We proposed to refine methods of palpating the trachea that we studied in previous experiments. We found that palpation of the anterior trachea with the fingertips during intubation enabled us to feel the tip of the endotracheal tube sliding into the trachea and improve correct depth compared to measurement at the teeth. 15 That study was undertaken to determine whether palpation of the trachea could enable correct position of the endotracheal tube with respect to depth. Esophageal intubation was studied subsequently, but the study was stopped when it became clear that we could not determine esophageal intubation by anterior tracheal palpation (unpublished).

However, during two instances of inadvertent esophageal intubation, we accidentally discovered a technique that may be able to detect inadvertent esophageal intubation as well as ensure correct endotracheal tube depth. Following tracheal intubation, with the cuff inflated to 50cm water pressure in the trachea, there was a sudden marked increase in the force necessary to gently tug the endotracheal tube proximally as the inflated cuff impinges on the rigid, encircling cricoid cartilage. When the increased force is sensed, then pushing the ETT down 2cm will ensure it is correctly positioned. If the cuff is in the esophagus, it will slide out without the sudden increased force being felt.

We plan a clinical pilot study of intubation of esophagus versus trachea with initial intubation of the esophagus flowed by intubation of the trachea.

Hypotheses. The force required for esophageal extubation with cuff inflated will be that required for tracheal extubation.

Primary outcome. To assess the reliability and accuracy of TETT as a method to determine tracheal versus esophageal intubation by measuring the force needed to slowly pull the ETT from the esophagus versus from the trachea.

Secondary outcomes. To find the optimal cuff-inflation pressure to distinguish trachea from esophagus and to assess the reliability and accuracy of TETT as a method to determine depth of endotracheal tube in the trachea.

Experimental design. A clinical trial with an objective measure of the difference in force of tugging between esophagus and trachea.

Patient safety. Intentional esophageal intubation has been reported in three previous airway studies with no harm coming to 275 patients. 16-18 Intentional intubation of the esophagus has been practiced routinely for gastroscopy in millions of patients. Mortality attributable to esophageal endoscopy is exceedingly low (0.005-0.01%), includes very sick patients, and occurs only with interventions such as biopsy and cautery of esophageal varices.19 In a prospective study of resident trainees performing upper G.I. endoscopy (N = 4,490), there were no complications attributable to insertion of the gastroscope in the upper third of the esophagus.20 The manoeuvre takes only about 10 seconds, then the opposite orifice can be intubated, with mask oxygenation between intubations if indicated. In a just-completed study of moving and ETT upward in the trachea with the cuff inflated to 50cm H2O pressure we found no increase in sore throat as a surrogate for tracheal damage in patients who had the ETT moved with cuff inflated compared to standard care (manuscript in preparation). 21 A recent study conducted at University of Saskatchewan showed that there is great variance in cuff inflation pressures clinically (manuscript in preparation), with pressures often exceeding 120 cm H2O pressure with no apparent adverse effects for inflation during surgery.

Clinical Utility. If this technique proves reliable, it can decrease the risk of ETT misplacement. Further, if it is reliable, it is particularly useful because it takes no special equipment, can be performed in less than 10 seconds anywhere from operating room to battlefield, and may make xray confirmation of ETT depth unnecessary, avoiding radiation and expense.

Methods

Participants:

1. Patients: Following University of Saskatchewan Research Ethics Board and Saskatoon Health Region approval, informed consent will be obtained from 20 patient participants. The collection, use and disclosure of patients' private information will conform to the Health Information Protection Act (HIPA). A convenience sample of American Society of Anesthesiologists (ASA) Class I and II patients ≥18 years, undergoing elective surgical procedures in the Saskatoon acute care hospitals of the Saskatoon Health Region and requiring endotracheal intubation as a component of the anesthetic plan, will be recruited. 22 Recruitment will take place in the Pre-Admission Clinic (PAC); in the Same Day Surgery and Day Surgery admission areas; and in the Operating Room (OR) Holding Area. Excluded patients will be those who are physiologically unstable, if there is urgency to proceed with surgery, patients requiring rapid sequence induction, and those with respiratory distress. The anesthesiologists will be encouraged to exclude patients if for any reason they feel that inclusion puts them at risk.
2. Testers: we will recruit and explain the manoeuvre to willing anesthesia staff, residents, and anesthesia assistants.

Interventions: Intubation will be by the attending anesthesiologist, who will choose the intubating anesthetic and equipment on clinical grounds. The anesthesiologists will intubate the esophagus first, and inflate the ETT cuff to their customary pressure, which we will then measure. An apparatus including a force transducer (LoadStar F-152217557 S-beam sensor run on LoadVue software; Loadstar Sensors Ltd., Fremont CA, USA) will be attached to the ETT connector and the testers will perform the gentle tugging while recording the force of pull until the ETT comes out of the esophagus. The process will be repeated with the trachea. At this point the anesthesiologist will intubate the trachea and proceed with surgical anesthesia. Only one set of intubations will be tested on any participant.

Measurements: Data will be recorded on paper data sheets for later transcription to a computer spread sheet for analysis. Usual demographics (age, gender, height, weight, type of surgery) will be recorded. Force transducer data will be digitally recorded on a computer for later analysis.

Sample size. Assuming that the anesthesiologist is able to intubate the esophagus successfully 100% of the time in this population, and the palpation technique is able to detect the esophageal intubation correctly only 50% of the time, we will need 15 participants assuming an alpha value of 0.05 and a beta value of 0.2 with Yates correction. Therefore, accounting for unforeseen exigencies, we will plan to recruit 20 participants.

Statistical Analysis: Demographics will be reported. Forces will be compared with paired t-tests.

Table 1. Diagnosis of esophageal intubation. Test ↓ Truth → T E totals T E totals

We will plot and subtract the force change from esophagus from the force change from trachea at the various pressures and construct a receiver operating curve to show the optimal cuff inflation pressure.

References

1. Caplan RA, Posner KL, Ward RJ, Cheney FW. Adverse respiratory events in anesthesia: a closed claims analysis. Anesthesiology 1990; 72: 828-33.
2. Schwartz DE, Matthay MA, Cohen NH. Death and other complications of emergency airway management in critically ill adults. A prospective investigation of 297 tracheal intubations. Anesthesiology 1995; 82: 367-76.
3. Clyburn P, Rosen M. Accidental oesophageal intubation. BrJ Anaesth 1994; 73: 55-63.
4. Harris EA, Arheart KL, Penning DH. Endotracheal tube malposition within the pediatric population: a common event despite clinical evidence of correct placement. Can J Anaesth 2008; 55: 685-90.
5. Owen RL, Cheney FW. Endobronchial intubation: a preventable complication. Anesthesiology 1987; 67: 255-7.
6. Mackenzie M, MacLeod K. Repeated inadvertent endobronchial intubation during laparoscopy. BrJ Anaesth 2003; 91: 297-8.
7. Evron S, Weisenberg M, Harow E, et al. Proper insertion depth of endotracheal tubes in adults by topographic landmarks measurements. J ClinAnesth 2007; 19: 15-9.
8. Ledrick D, Plewa M, Casey K, Taylor J, Buderer N. Evaluation of manual cuff palpation to confirm proper endotracheal tube depth. PrehospDisasterMed 2008; 23: 270-4.
9. Pattnaik SK, Bodra R. Ballotability of cuff to confirm the correct intratracheal position of the endotracheal tube in the intensive care unit. EurJ Anaesthesiol 2000; 17: 587-90.
10. Pollard RJ, Lobato EB. Endotracheal tube location verified reliably by cuff palpation. Anesth Analg 1995; 81: 135-8.
11. Muslu B, Sert H, Kaya A, et al. Use of sonography for rapid identification of esophageal and tracheal intubations in adult patients. Journal of ultrasound in medicine : official journal of the American Institute of Ultrasound in Medicine 2011; 30: 671-6.
12. McKay WP, Wang A, Yip K, Raazi M. Tracheal ultrasound to assess endotracheal tube depth: an exploratory study. CanJAnaesth 2015.
13. Hoffmann B, Gullett JP, Hill HF, et al. Bedside ultrasound of the neck confirms endotracheal tube position in emergency intubations. Ultraschall in der Medizin (Stuttgart, Germany : 1980) 2014; 35: 451-8.
14. Ramsingh D, Frank E, Haughton R, et al. Auscultation versus Point-of-care Ultrasound to Determine Endotracheal versus Bronchial Intubation: A Diagnostic Accuracy Study. Anesthesiology 2016; 124: 1012-20.
15. McKay WP, Klonarakis J, Pelivanov V, O'Brien JM, Plewes C. Tracheal palpation to assess endotracheal tube depth: an exploratory study. Canadian journal of anaesthesia = Journal canadien d'anesthesie 2014; 61: 229-34.
16. Sharieff GQ, Rodarte A, Wilton N, Silva PD, Bleyle D. The self-inflating bulb as an esophageal detector device in children weighing more than twenty kilograms: a comparison of two techniques. Annals of emergency medicine 2003; 41: 623-9.
17. Tong YL, Sun M, Tang WH, Xia JY. The tracheal detecting-bulb: a new device to distinguish tracheal from esophageal intubation. Acta anaesthesiologica Sinica 2002; 40: 159-63.
18. Zaleski L, Abello D, Gold MI. The esophageal detector device. Does it work? Anesthesiology 1993; 79: 244-7.
19. Schrag SP, Sharma R, Jaik NP, et al. Complications related to percutaneous endoscopic gastrostomy (PEG) tubes. A comprehensive clinical review. J GastrointestinLiver Dis 2007; 16: 407-18.
20. Schauer PR, Schwesinger WH, Page CP, Stewart RM, Levine BA, Sirinek KR. Complications of surgical endoscopy. A decade of experience from a surgical residency training program. SurgEndosc 1997; 11: 8-11.
21. Liu J, Zhang X, Gong W, et al. Correlations between controlled endotracheal tube cuff pressure and postprocedural complications: a multicenter study. Anesthesia and analgesia 2010; 111: 1133-7.
22. Saubermann AJ, Lagasse RS. Prediction of rate and severity of adverse perioperative outcomes: "normal accidents" revisited. The Mount Sinai journal of medicine, New York 2012; 79: 46-55.

ELIGIBILITY:
Inclusion Criteria: American Society of Anesthesiologists (ASA) Class I and II patients ≥18 years, undergoing elective surgical procedures in the Saskatoon acute care hospitals of the Saskatoon Health Region and requiring endotracheal intubation as a component of the anesthetic plan -

Exclusion Criteria: those who are physiologically unstable, if there is urgency to proceed with surgery, patients requiring rapid sequence induction, and those with respiratory distress. The anesthesiologists will be encouraged to exclude patients if for any reason they feel that inclusion puts them at risk.

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P McKay, MD, Principal Investigator — University of Saskatchewan Dept. of Anesthesiology
Locations (1):
- Saskatoon Health Region, 410 22nd Street East, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intubated Patient: Esophagus, then trachea, are intentionally intubated with a cuffed endotracheal tube, the cuff inflated to >30cm water pressure, a force transducer attached, and force of extubation recorded.
Period: Overall Study
Arm/Group | Intubated Patient
Started | 11
Completed | 10
Not Completed | 1
Not completed — Force transducer technical failure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esophageal Then Tracheal Intubated Patient
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] — years
  years | 61 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
height [Mean (Standard Deviation); unit: cm] — cm
  cm | 170 (9)
weight [Mean (Standard Deviation); unit: kg] — kg
  kg | 80 (19)

OUTCOME MEASURES:

1. Primary Outcome: Withdrawal Force.
Description: Force (N) of resistance to pulling the tube out compared for esophageal versus tracheal intubation
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Newtons
Groups:
- Esophagus: withdrawal force (N)
Arm/Group | Esophagus
Number analyzed (Participants) | 11
Newtons
  esophagus | 6.2 (4.4)
  trachea | 6.1 (2.0)
Statistical Analysis 1: Comparison: Esophagus; Test type: Superiority; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-2.4 to 2.6], Standard Deviation 4.4

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Intubated Patient: all participants
Arm/Group | Intubated Patient
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03480425/Prot_SAP_000.pdf